CLINICAL TRIAL: NCT01450033
Title: A Peer Mentoring Intervention to Improve Adherence and Quality of Life in Adolescents With Solid Organ Transplants
Brief Title: Peers for Promoting Adolescent Transplant Health
Acronym: Peers4PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-008336; DK083529 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: kidney; renal; transplant; transplantation; adolescent; pediatric; mentor; mentoring; medication; adherence; immunosuppressant; heart; liver
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Standard of care
- Mentoring group (Experimental): Subjects in this group will participate in the following intervention activities: medical record review; questionnaires including the Hollingshead Socioeconomic Status Survey, modified Medication Adherence Module, Peds QL Transplant Module, Medical Outcomes Study Social Support Scale, and self-efficacy scale; in-person meetings with mentor; e-communication with mentor (i.e. texts, Facebook, phone calls, etc); and collection of pharmacy refill data and clinical data.
  Interventions: Behavioral: Peer Mentoring; Behavioral: e-Communication with mentor

INTERVENTIONS:
Behavioral: Peer Mentoring — Subjects will be assigned a peer mentor who will provide social support primarily via e-communication. They will also meet in-person at study entry, 6 months and 1-year.
  Arms: Mentoring group
Behavioral: e-Communication with mentor — Subjects will interact on a mutually agreeable basis via their choice of text messaging, Facebook, phone calls, emails, and other formats
  Arms: Mentoring group

SUMMARY:
Adolescents with solid organ transplants have poorer outcomes than adults, and do not respond as well to post-rejection treatment. In addition to well-recognized declines in individual health-related quality of life, premature graft loss creates considerable health and economic burdens. High nonadherence rates among adolescents are believed to contribute majorly to rejection, premature allograft dysfunction and failure. Studies suggest that a telephone-based peer mentoring approach, with texting and e-communication, is a promising, practical means to promote medication adherence in adolescent solid organ transplant recipients. The study's main objectives are 1) to determine the efficacy of peer mentoring to improve medication adherence and health-related quality of life vs. usual care in adolescents and young adults with solid organ transplants, and 2) to determine the mechanisms through which peer mentoring impacts medication adherence and health-related quality of life.

DETAILED DESCRIPTION:
The investigators will conduct a single-center Phase II randomized clinical trial in which adolescents ages 14-23 and greater 3 months post solid organ transplant will receive either a peer mentor or usual care. The investigators will assess changes in quality of life from baseline to one year post-study entry. The investigators will also examine adherence changes over the same time frame using pharmacy refill data and a questionnaire. Peer mentors will provide social support and promote subject self-efficacy primarily via e-communication. Changes in social support and self-efficacy will be measured over a one-year period.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 14 to 23 years
* Greater than one year post kidney, heart or liver transplant
* Able to speak and read in English
* Willing and able to provide informed consent or assent
* Parental guardian permission (informed consent) if appropriate

Exclusion Criteria:

* Unwilling to participate
* Unable to speak or read in English
* Unable to provide informed assent or consent
* Estimated glomerular filtration rate (eGFR) less than 20 ml/min/1.73m^2
* On dialysis
* Less than three months post transplant
* Post-transplant lymphoproliferative disease

Ages: 14 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2011-09; Primary Completion 2017-01 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 1 year
  The primary endpoint is medication adherence, defined by the modified Medication Adherence Module (MAM), standard deviations of immunosuppressive drug levels, percent adherence from pharmacy refill data and pill counts at 1 year.

SECONDARY OUTCOMES:
Mentoring mechanisms | 1 year
  The secondary endpoint is to determine the mechanisms through which peer mentoring impacts medication adherence and healthcare-related quality of life. It is hypothesized that peer mentors will provide social support which will improve subject self-efficacy.
Quality of Life | 1 year
  Health-related Quality of Life (QL) will be measured using the Peds QL Transplant Module.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Amaral, MD, MHS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829